CLINICAL TRIAL: NCT00576160
Title: Improving Med Adherence in Post-ACS Patients: Phase 1B Dose-Finding RCT
Brief Title: Improving Medication Adherence in Post-ACS Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This was a dosing study to determine acceptability. Participants found protocol burdensome and so we terminated.
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Karina Davidson, Professor of Medicine in Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAB9215; K24HL084034 (NIH)
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Medication Adherence; Acute Coronary Syndrome
Keywords: medication adherence
MeSH Terms: conditions — Medication Adherence; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Participants will complete Baseline and 30-day assessment visit. At both visits BDI II, Self-Efficacy Questions, AEs Assessment, and Treatment Satisfaction will be assessed. A MEMS cap will be used during the 30-day period to asses medication adherence to their prescribed aspirin.
  Usual Care: Participants assigned to UCC will only receive the pre- and post-assessment session, and any adherence education or encouragement that is regularly provided by their treating physicians.
- B (Experimental): Participants will complete Baseline and 30-day assessment visit. At both visits BDI II, Self-Efficacy Questions, AEs Assessment, and Treatment Satisfaction will be assessed. A MEMS cap will be used during the 30-day period to asses medication adherence to their prescribed aspirin. After Baseline, there is an initial session telephone session with PST therapist. Subsequent treatment sessions provide a context for the patient to discuss the problems and difficulties they face and that give rise to medication non-adherence.
  Interventions: Behavioral: PST therapy

INTERVENTIONS:
Behavioral: PST therapy — Problem-Solving Therapy (PST) is a behavioral approach that teaches patients how to systematically solve their own behavioral difficulties. During telephone treatment sessions, the patient will discuss the problems and difficulties they face and that give rise to medication non-adherence.
  Arms: B

SUMMARY:
Many post Acute Coronary Syndrome(ACS) patients do not take their medications (including aspirin) as prescribed, leading to an increase in mortality. Patients enrolled in this study will be enrolled into one of two groups. Patients in the first group will have their medication adherence measured, but will receive all other care as usual. Patients in the second group will also have their medication adherence measured, but they will receive telephone-delivered problem solving therapy (PST) in addition to their usual care. The two groups will be combined to determine the Minimally Effective Dose (MED) and the Maximally Tolerated Dose (MTD) for adherence to aspirin. The medication adherence of the PST group will improve by 20% (<55% to >75%).

ELIGIBILITY:
Inclusion Criteria:

1. Medical eligibility:

   1. Patient presenting for staged intervention with positive cardiac history OR
   2. Patient with stable CAD who received cardiac admission but does not report chest pain. OR
   3. Patient with stable CAD who has had a cardiac admission in the past.
2. Patient is non-adherent to prescribed medication.

The following exclusion criteria have been set for either safety concerns or concerns that patients will not be able to complete the protocol:

1. inability to communicate in English or Spanish
2. unwilling to be randomized or to have aspirin in a separate bottle if they use a pill box
3. unavailability for the 1 month period of the study (including being unavailable by phone and/or traveling out of the country)
4. medically unable to receive aspirin (e.g. allergy, contra-indicated, etc)
5. deemed unable to comply with the protocol (either self selected or by indicating during screening that s/he could not complete all requested tasks). This includes patients with a level of cognitive impairment indicative of dementia, and patients with current alcohol or substance abuse.
6. deemed to need immediate psychiatric assessment (e.g., must be hospitalized, or have some other psychiatric intervention conducted within 72 hours).
7. active psychosis, bipolar disorder, or any overt personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of medication adherence | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Karina W. Davidson, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States